CLINICAL TRIAL: NCT05541497
Title: Varenicline for Treatment of E-cigarette Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000032740; 000 (Other: CTGTY)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Smoking Cessation
Keywords: e-cigarette
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Varenicline + Self-Change Pamphlet (Experimental): * Days 1-3: 0.5mg study pill once per day
  * Days 4-7: 0.5mg study pill twice per day
  * Weeks 2-8: 1mg study pill twice per day in combination with a minimal, self-guided behavior change booklet. This booklet includes general tips for e-cigarettes cessation and information about the free web-based e-cigarette cessation program sponsored by The Truth Initiative and Mayo called "This is Quitting". This study will have an 8-week treatment period and a 4-week follow-up.
  Interventions: Drug: Varenicline Tartrate
- Placebo + Self-Change Pamphlet (Placebo Comparator): * Days 1-3: 0.5mg placebo pill once per day
  * Days 4-7: 0.5mg placebo pill twice per day
  * Weeks 2-8: 1mg placebo pill twice per day in combination with a minimal, self-guided behavior change booklet. This booklet includes general tips for e-cigarettes cessation and information about the free web-based e-cigarette cessation program sponsored by The Truth Initiative and Mayo called "This is Quitting". This study will have an 8-week treatment period and a 4-week follow-up.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline Tartrate — Days 1-3: 0.5mg study pill once per day, Days 4-7: 0.5mg study pill twice per day, Weeks 2-8: 1mg study pill twice per day
  Arms: Varenicline + Self-Change Pamphlet
Drug: Placebo — Days 1-3: 0.5mg pill once per day, Days 4-7: 0.5mg pill twice per day, Weeks 2-8: 1mg pill twice per day
  Arms: Placebo + Self-Change Pamphlet

SUMMARY:
Varenicline is used to treat tobacco use dependence. It helps reduce cravings for tobacco use and decreases the pleasurable effects of cigarettes and other tobacco products. Varenicline has been proven to reduce the desire to smoke cigarettes. This study aims to test whether it shows a similar benefit for individuals who vape and are interested in quitting.

DETAILED DESCRIPTION:
Varenicline is a highly efficacious FDA-approved smoking cessation pharmacotherapy. The aim of this study is to examine the effectiveness of varenicline for e-cigarette cessation medication for mono- e-cigarette use in combination with a minimal, self-guided behavior change booklet. This booklet will include general tips for e-cigarettes cessation and information about the free web-based e-cigarette cessation program sponsored by The Truth Initiative and Mayo called "This is Quitting". This study will have an 8-week treatment period and a 4-week follow-up phase. Participants will be randomized to receive an 8-week supply of varenicline or matching placebo (gel capsule filled with cellulose powder) in combination with the self-change booklet. The investigators hypothesize that participants who receive varenicline will have higher rates of e-cigarette cessation.

ELIGIBILITY:
Inclusion Criteria:

* daily use of an e-cigarette containing nicotine (defined as use for at least 25 days out of the past month)
* use of an e-cigarette containing nicotine> 6 months
* have desire to quit e-cigarettes, are willing to set a quit date and maintain e-cigarette abstinence
* have daily access to a smartphone or have regular (daily) access/use of email
* live in South Carolina or Connecticut

Exclusion Criteria:

* Vulnerable Populations: Not be enrolling vulnerable populations, specifically pregnant women, children, prisoners, or institutionalized individuals
* The investigators will not enroll participants incapable of providing their own consent. The rationale will be provided to the individual as well as his or her family members.

Referrals for further evaluation, including urgent or emergent evaluation, will be made as needed and clinically warranted.

* exclude individuals with medical contraindications for varenicline use (i.e., severe renal impairment)
* exclude anyone currently using smoking cessation medications.
* Individuals will also be excluded if another household member is currently enrolled in the study.
* Individuals will be excluded if not proficient in English.
* Individuals will be excluded if they have smoked any combustible cigarettes in the past 6 months.
* Verification of Non-Pregnancy: Females ages <55 will be mailed a commercially available pregnancy test to verify non-pregnancy. Written confirmation of negative pregnancy test via REDCap will be required prior to enrollment in the trial. Participants are also informed that they should let us know if they become pregnant during the trial. Medications will not be sent until this verification is in place. These procedures are based on the Medical University of South Carolina Internal Review Board approved STARS protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fucito, Ph.D., Principal Investigator — Yale University; Benjamin Toll, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline + Self-Change Pamphlet: * Days 1-3: 0.5mg study pill once per day
  * Days 4-7: 0.5mg study pill twice per day
  * Weeks 2-8: 1mg study pill twice per day in combination with a minimal, self-guided behavior change booklet. This booklet includes general tips for e-cigarettes cessation and information about the free web-based e-cigarette cessation program sponsored by The Truth Initiative and Mayo called "This is Quitting". This study will have an 8-week treatment period and a 4-week follow-up.
  Varenicline Tartrate: Days 1-3: 0.5mg study pill once per day, Days 4-7: 0.5mg study pill twice per day, Weeks 2-8: 1mg study pill twice per day
- Placebo + Self-Change Pamphlet: * Days 1-3: 0.5mg placebo pill once per day
  * Days 4-7: 0.5mg placebo pill twice per day
  * Weeks 2-8: 1mg placebo pill twice per day in combination with a minimal, self-guided behavior change booklet. This booklet includes general tips for e-cigarettes cessation and information about the free web-based e-cigarette cessation program sponsored by The Truth Initiative and Mayo called "This is Quitting". This study will have an 8-week treatment period and a 4-week follow-up.
  Placebo: Days 1-3: 0.5mg pill once per day, Days 4-7: 0.5mg pill twice per day, Weeks 2-8: 1mg pill twice per day
Period: Overall Study
Arm/Group | Varenicline + Self-Change Pamphlet | Placebo + Self-Change Pamphlet
Started | 20 | 20
Completed 8 Weeks of Treatment | 18 | 17
Completed 12 Week Follow up | 18 | 15
Completed | 18 | 15
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline + Self-Change Pamphlet | Placebo + Self-Change Pamphlet | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (10.3) | 28.1 (6.4) | 28.2 (8.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 10 | 10 | 20
  Female | 9 | 10 | 19
  Transgender | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
History of smoking [Count of Participants; unit: Participants] | 10 | 11 | 21
Vaping Continuously All Day [Count of Participants; unit: Participants] | 15 | 18 | 33
Years of E-cigarette Use [Mean (Standard Deviation); unit: years] | 4.9 (2.8) | 4.8 (1.8) | 4.9 (2.4)
E-cigarette Dependence [Mean (Standard Deviation); unit: score on a scale] — Dependence assessed by standardized Patient-Reported Outcomes Measurement System (PROMIS) 4-item measure.Total score range 4-20. Higher scores indicate more dependence.
  score on a scale | 13.4 (3.6) | 15 (2.8) | 14.2 (3.3)
Type of E-cigarette Devices Used [Number; unit: device]
  Disposable | 8 | 12 | 20
  Closed Pod/Cartridge | 9 | 5 | 14
  Refillable Pod/Cartridge | 1 | 3 | 4
  Refillable Tank | 2 | 0 | 2
Nicotine Salt-Based E-Cigarette [Count of Participants; unit: Participants] | 17 | 19 | 36
Comorbid Conditions [Count of Participants; unit: Participants]
  Any | 9 | 7 | 16
  Depression | 6 | 3 | 9
  Anxiety | 6 | 4 | 10
  Other psychiatric | 5 | 1 | 6
  Other substance use disorder | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Abstinent From Vaping at Week 8
Description: Abstinence is defined as no vaping, not even a puff, every day for the last 7 days via self-report (i.e., 7 day point prevalent abstinence).
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Self-Change Pamphlet | Placebo + Self-Change Pamphlet
Number analyzed (Participants) | 20 | 20
Participants | 9 | 6
Statistical Analysis 1: Comparison: Varenicline + Self-Change Pamphlet vs Placebo + Self-Change Pamphlet; Test type: Superiority; Risk Ratio (RR) = 1.51, 95% CI 2-sided [0.68 to 3.37]

2. Secondary Outcome: Number of Participants Abstinent From Vaping at Week 12
Description: as for outcome 1
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Self-Change Pamphlet | Placebo + Self-Change Pamphlet
Number analyzed (Participants) | 20 | 20
Participants | 8 | 6
Statistical Analysis 1: Comparison: Varenicline + Self-Change Pamphlet vs Placebo + Self-Change Pamphlet; Test type: Superiority; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.59 to 3.13]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Varenicline + Self-Change Pamphlet | Placebo + Self-Change Pamphlet
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 12/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline + Self-Change Pamphlet (N=20) | Placebo + Self-Change Pamphlet (N=20)
Headache (Nervous system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 4 | 1 — Vivid Dreams
Depressed Mood (Psychiatric disorders) | 1 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 — Lightheadedness
Irritability (Psychiatric disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 — Stomach ache
Insomnia (Psychiatric disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 — Appetite Changes
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 — Indigestion
Belching (Gastrointestinal disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT05541497/Prot_SAP_000.pdf